CLINICAL TRIAL: NCT00124579
Title: S0417 A Phase II Study of Bortezomib (Velcade™, PS-341), Thalidomide, and Dexamethasone in Patients With Refractory Multiple Myeloma
Brief Title: S0417 Bortezomib, Thalidomide, and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0417; S0417 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Multiple Myeloma
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bortezomib with thalidomide and dexamethasone (Experimental): bortezomib with thalidomide and dexamethasone
  Interventions: Drug: bortezomib; Drug: dexamethasone; Drug: thalidomide

INTERVENTIONS:
Drug: bortezomib — induction: 1 mg/m2 IV push days 1, 4, 8, 11 every 21 days
Drug: dexamethasone — induction: 20 mg/d PO days 1, 2, 4, 5, 8, 9, 11, 12 every 21 days maintenance: 40 mg days 1-4 every 28 days until progression
Drug: thalidomide — 100 mg/d PO days 1-21 every 21 days

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as thalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. It may also stop the growth of cancer by blocking blood flow to the cancer. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with thalidomide and dexamethasone may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with thalidomide and dexamethasone works in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the confirmed overall response rate (complete remission, remission, and partial remission) in patients with relapsed or refractory multiple myeloma treated with bortezomib, thalidomide, and dexamethasone.
* Determine overall and progression-free survival of patients treated with this regimen.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Correlate, preliminarily, treatment with bortezomib with the activation of osteoblasts in these patients.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive bortezomib IV on days 1, 4, 8, and 11, oral thalidomide once daily on days 1-21, and oral dexamethasone once daily on days 1, 2, 4, 5, 8, 9, 11, and 12. Treatment repeats every 21 days until achievement of confirmed complete remission (CR), remission (R), or partial remission (PR) OR for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients achieving confirmed CR, R, or PR who reach a plateau prior to receiving the maximum 8 courses of induction therapy OR who achieve confirmed CR, R, or PR after receiving the maximum 8 courses of induction therapy proceed to maintenance therapy. Patients achieving stable disease after receiving the maximum 8 courses of induction therapy either proceed to maintenance therapy or receive further treatment with bortezomib, thalidomide, and dexamethasone off-study.

* Maintenance therapy: Patients receive oral dexamethasone on days 1-4. Courses repeat every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed within 30 days and then every 6 months for up to 5 years.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma (MM)

  * Active disease
* Relapsed or refractory disease after ≥ 1 prior therapy for MM, that may have included autologous or allogeneic stem cell transplantation

  * Relapse is defined as the occurrence of any of the following during or after prior treatment:

    * Myeloma protein level increase by > 100% from the lowest previously recorded level
    * Myeloma protein level increase above the defined response criteria for partial remission
    * Reappearance of any myeloma peak that had disappeared during the prior treatment
    * Increase in the size and number of lytic bone lesions and/or focal lesions by x-ray, MRI, positron emission tomography, and/or CT scan
  * Refractory disease is defined as no response (i.e., not achieving complete remission, remission, or partial remission) to prior therapy
* Measurable disease
* No evidence of POEMS (polyneuropathy, organomegaly, endocrinopathy, presence of M-protein, and skin changes) syndrome
* Must be registered on protocol SWOG-S0334

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2 (unless due to bone pain)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 50,000/mm^3

Hepatic

* AST or ALT ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 3 times ULN

Renal

* Creatinine clearance > 30 mL/min

Cardiovascular

* No New York Heart Association class III or IV congestive heart failure
* No myocardial infarction within the past 6 months
* No poorly controlled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective double method contraception for ≥ 4 weeks before, during, and for ≥ 4 weeks after completion of study treatment (during and for 4 weeks after completion of study treatment for male patients)
* No blood, ova, or sperm donation during study treatment
* No active infection requiring antibiotics
* No neurotoxicity ≥ grade 2
* No diabetes mellitus
* No other serious medical or psychiatric illness that would preclude study treatment
* No other malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* At least 14 days since prior chemotherapy (28 days for nitrosoureas) and recovered

Endocrine therapy

* Not specified

Radiotherapy

* At least 14 days since prior radiotherapy and recovered

Surgery

* Not specified

Other

* No prior bortezomib alone or combined with thalidomide
* Concurrent participation on protocol SWOG-S0309 allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-08; Primary Completion 2008-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordan Srkalovic, MD, PhD, Principal Investigator — Sparrow Regional Cancer Center; Mohamad A. Hussein, MD, Principal Investigator — The Cleveland Clinic
Locations (127):
- United States (127):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Foote Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Center for Cancer Medicine and Blood Disorders, PA, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib With Thalidomide and Dexamethasone Induction: Induction (per 21-day cycle): Bortezomib - 1.0 mg/m2 (Days 1, 4, 8, and 11). Dexamethasone - 20 mg/d PO (Days 1, 2, 4, 5, 8, 9, 11, and 12). Thalidomide 100 mg (Days 1-21).
  Maintenance (per 28-day cycle): thalidomide 100mg (Days 1-28). Dexamethasone 40 mg Days 1-4.
Period: Induction
Arm/Group | Bortezomib With Thalidomide and Dexamethasone Induction
Started | 7
Completed | 2
Not Completed | 5
Period: Maintenance
Arm/Group | Bortezomib With Thalidomide and Dexamethasone Induction
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Bortezomib With Thalidomide and Dexamethasone: Induction (per 21-day cycle): Bortezomib - 1.0 mg/m2 (Days 1, 4, 8, and 11). Dexamethasone - 20 mg/d PO (Days 1, 2, 4, 5, 8, 9, 11, and 12). Thalidomide 100 mg (Days 1-21).
  Maintenance (per 28-day cycle): thalidomide 100mg (Days 1-28). Dexamethasone 40 mg Days 1-4.
Arm/Group | Bortezomib With Thalidomide and Dexamethasone
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 63.7 [37.6 to 81.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3

OUTCOME MEASURES:

1. Secondary Outcome: Toxicity Evaluation
Description: To evaluate the qualitative and quantitative toxicities associated with this regimen.
Time Frame: From date of protocol therapy start to date of protocol therapy end, i.e., up to about 3.5 years
Population: All participants receiving at least one dose of induction therapy
Measure: Number; unit: Participants
Groups:
- Bortezomib + Thal/Dex: Induction (per 21-day cycle): Bortezomib - 1.0 mg/m2 (Days 1, 4, 8, and 11). Dexamethasone - 20 mg/d PO (Days 1, 2, 4, 5, 8, 9, 11, and 12). Thalidomide 100 mg (Days 1-21).
  Maintenance (per 28-day cycle): thalidomide 100mg (Days 1-28). Dexamethasone 40 mg Days 1-4.
Arm/Group | Bortezomib + Thal/Dex
Number analyzed (Participants) | 7
Participants
  Albumin, serum-low (hypoalbuminemia) | 1
  Allergy/Immunology-Other | 1
  Bilirubin (hyperbilirubinemia) | 1
  Edema: limb | 1
  Extremity-lower (gait/walking) | 1
  Fatigue (asthenia, lethargy, malaise) | 1
  Hemoglobin | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 1
  Leukocytes (total WBC) | 1
  Lymphopenia | 1
  Muscle weakness, not d/t neuropathy - Extrem-lower | 1
  Muscle weakness, not d/t neuropathy - body/general | 1
  Neuropathy: motor | 1
  Neuropathy: sensory | 1
  Neutrophils/granulocytes (ANC/AGC) | 2
  Platelets | 1

2. Primary Outcome: Overall Response Rate Complete Remission (CR), Remission (R), and Partial Remission (PR).
Description: Responses are defined as follows:
  Complete Remission: Absence of bone marrow or blood findings of multiple myeloma. This includes disappearance of all evidence of serum and urine M-proteins on immunofixation electrophoresis studies. Normalization of serum concentrations of normal immunoglobulins is not required for CR. There must also be no evidence of increasing anemia. Bone marrow cellularity must be ≥ 20% with plasma cells ≤ 5%.
  Remission: A ≥ 75% reduction in the serum M-protein, and if a urine M-protein (Bence-Jones protein) is present, either a ≥ 90% reduction in this protein, or a urine M-protein < 0.2gm/day. Bone marrow plasma cells must be ≤ 5%.
  Partial Remission: A ≥ 50% reduction in the serum M-protein, and if present, a ≥ 50% reduction in the urine M-protein (Bence-Jones protein). Bone marrow plasma cells must not be increased from baseline level.
Time Frame: 1 year
Population: Ninety patients is sufficient to distinguish between the null hypothesis that the response rate is 45% versus the alternative of a response rate of 60% with 89% power, using a one-sided test based on the binomial distribution with a significance level of 5%.
Measure: Number; unit: percentage of participants
Arm/Group | Bortezomib With Thalidomide and Dexamethasone
Number analyzed (Participants) | 7
percentage of participants | 14

3. Secondary Outcome: Progression-Free Survival
Description: From date of initial registration to date of progression/relapse of disease (> 25% increase from baseline in myeloma protein production or other signs of disease progression such as hypercalcemia, etc.) or death from any cause, whichever came first, up to 5 years
Time Frame: about 12-18 months
Population: With ninety patients, we will have 82% power to rule out a null hypothesis of a 12-month median survival versus an alternative hypothesis of an 18-month median survival at a significance level of 5%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bortezomib With Thalidomide and Dexamethasone
Number analyzed (Participants) | 7
Months | 8 [4 to 12]

ADVERSE EVENTS:
Arm/Group | Bortezomib + Thal/Dex
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Thal/Dex (N=7)
Edema: limb (General disorders) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Platelets (Investigations) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Thal/Dex (N=7)
Hemoglobin (Blood and lymphatic system disorders) | 6
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1
SVT and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 1
Cushingoid appearance (Endocrine disorders) | 1
Night blindness (nyctalopia) (Eye disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Watery eye (epiphora, tearing) (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 1
Distention/bloating, abdominal (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Edema: head and neck (General disorders) | 1
Edema: limb (General disorders) | 3
Extremity-lower (gait/walking) (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 7
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 2
Pain-Other (General disorders) | 2
Rigors/chills (General disorders) | 1
Allergy/Immunology-Other (Immune system disorders) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Bladder (Infections and infestations) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Soft tiss (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 1
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 1
Infection-Other (Infections and infestations) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2
AST, SGOT (Investigations) | 1
Alkaline phosphatase (Investigations) | 2
Bilirubin (hyperbilirubinemia) (Investigations) | 2
Creatinine (Investigations) | 2
Leukocytes (total WBC) (Investigations) | 4
Lymphopenia (Investigations) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3
Platelets (Investigations) | 4
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 1
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2
Pain - Joint (Musculoskeletal and connective tissue disorders) | 2
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Neurology-Other (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 6
Pain - Head/headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mood alteration - depression (Psychiatric disorders) | 1
Glomerular filtration rate (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Sexual/Reproductive Function-Other (Specify) (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4
Hemorrhage, Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 1
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No